CLINICAL TRIAL: NCT04066127
Title: A Randomized Controlled Trial Comparing a New State-of-the-art Non Ischemic Heart Preservation Method With the Standard Ischemic Cold Static Storage Method of Donor Hearts in Adult Heart Transplantation
Brief Title: Non-ischaemic Heart Preservation Versus Standard Cold Storage in Human Heart Transplantation
Acronym: NIHP2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Johan Nilsson, MD, PhD, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018/941
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Transplant; Failure, Heart
Keywords: Heart preservation; Ex-vivo perfusion; Heart transplantation; Acute cellular rejection; Survival

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Acute cellular rejection assessment will be performed by a blinded access
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-ischemic heart preservation (NIHP) (Experimental): Non-ischemic hypothermic perfusion (NIHP): The donor heart is preserved using a portable heart-lung machine. The device perfuse the heart continuously with a a new preservation solution at a temperature of 8°C.
  Interventions: Device: Non-ischemic heart preservation (NIHP)
- Standard cold storage (SCS) (Other): Standard cold static storage (SCS): The donor heart is preserved using a standard crystalloid cardioplegia. The heart is in then storage i a transport box containing ice to keep the temperature around 4-8°C. The device does not perfuse the heart.
  Interventions: Device: Standard ischemic cold static storage (SCS)

INTERVENTIONS:
Device: Non-ischemic heart preservation (NIHP) — The device is a miniaturized and fully automated heart-lung machine, housed in a portable device (weight 32 kg), that enables transportation between hospitals. The reservoir is filled with 2.5 liters of the perfusion solution plus approximately 500 mL compatible washed and leucocyte-filtered red blood cells from the hospital blood bank. The NIHP system software is adjusted to maintain a mean blood pressure of 20-25 mmHg in the aortic root, giving a coronary flow between 150 mL/min and 250 mL/min.
  Arms: Non-ischemic heart preservation (NIHP)
Device: Standard ischemic cold static storage (SCS) — The device is a cool box that enables transportation between hospitals. The heart is stored on ice slush in the box at a temperature of approximately 4-8 °C.
  Arms: Standard cold storage (SCS)

SUMMARY:
The overall aim of this study is to compare a new state-of-the-art ex-vivo organ preservation method with standard ischemic cold static storage of donor hearts in adult cardiac transplantation.

Standard heart preservation before transplantation consists of cold ischemic storage of the heart. Clinical studies have shown that the morbidity and mortality risk increases with the extension of the allograft ischemic time over four hours. For each additional hour the mortality risk increase with 25% the first year. This time constraint is costly and results in severe logistical problems, leading to loss of transplantable organs. The preliminary results from our safety study, where six patients transplanted with the new state-of-the-art ex-vivo organ preservation method, have shown promising results.

The study is a multicenter, prospective, open, blinded endpoint, randomized, controlled clinical trial. The primary end-point is survival free of acute cellular rejection (ACR) and retransplantation within 1-year post-transplant. ACR will be assessed blinded. The secondary end-points are ischemia/reperfusion injury, early graft dysfunction, and QoL.

DETAILED DESCRIPTION:
SURVEY OF THE FIELD Ischemia and reperfusion (I/R) - elicited tissue injury contributes to morbidity and mortality. In organ transplantation, it is a major challenge. The imbalance in metabolic supply and demand within the ischemic organ results in tissue hypoxia and microvascular dysfunction. The following reperfusion enhances the activation of innate and adaptive immune responses resulting in a cell death program.

A damaged endothelium increases the risk of allograft rejection within 1-year after transplantation and a drug treated rejection increases the risk of chronicle rejection and five-year mortality. An improved preservation of the endothelium of the coronary arteries is therefore instrumental to achieve an improved short- and long-term outcome for the transplanted patients.

Standard heart preservation before transplantation consists of cold ischemic storage of the heart. Clinical studies have shown that the mortality risk increases sharply with extension of the allograft ischemic time over four hours. For each additional hour, the mortality risk increases with 25% the first year. Different myocardial cardioplegic preservation solutions and ex-vivo perfusion machines have been developed. Despite some promising experimental results, no consistent differences in outcome have been found. Our first-in-man pilot study, including 6 NIHP cases, show the device's feasibility and provide the first pieces of evidence that machines improves outcome of heart transplantation. However, as these results are based on a non-randomized study design with a few patients, a randomized study is needed to ensure the effect.

PURPOSE AND AIMS The purpose of this study is to compare a new state-of-the-art non ischemic heart preservation (NIHP) method, on heart allograft function, rejection episodes, and quality of life, with the standard ischemic cold static storage (SCS) method of donor hearts in adult heart transplantation.

STUDY DESIGN The study is a multicentre, prospective, randomized, open, blinded endpoint, controlled clinical trial. The study will randomly assign eligible patients to be transplanted with a donor heart preserved with either a new ex-vivo perfusion method (NIHP) or the standard cold static storage (SCS). The study will be performed at Skane University Hospital, Karolinska University Hospital, Linköping University Hospital, and Uppsala University Hospital, which cover two-thirds of the population in Sweden. Patients listed at these centres will be transplanted at Skane University Hospital and then returned to their centre for post-transplant care. The data collection, statistical analysis, and presentation of results will be done according to the CONSORT criteria. The main outcomes will be reported on intention to treat basis.

PICO Population: Adult patients with end-stage heart failure eligible for heart transplantation.

Intervention: Recipient transplanted with a donor heart preserved using NIHP. Control: Recipient transplanted with a donor heart preserved using SCS. Outcome: Survival, rejection, graft function, and quality-of-life.

STATISTICAL ANALYS PLAN Populations for analysis The full analysis set will consist of all randomized patients. Following the intent-to-treat principle, patients will be analyzed according to the preservation methods (NIHP and SCS, respectively) to which they were assigned at randomization. Efficacy variables will be analyzed based on all randomized patients as the primary population.

Patient demographics/other baseline characteristics Baseline value is defined as the last non-missing assessment prior to the transplantation. Summary statistics will be provided by treatment group for demographics and baseline characteristics, including age, sex, weight, height, body mass index (BMI), diagnosis, prior hospitalization, need for inotropic support pre-transplant and/or ECMO, CK-MB, TnI, proBNP, and vital signs. Continuous variables will be summarized using n, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized using frequency and percentage. The difference between treatment groups will be compared using the Chi-square test for categorical variables or using Mann-Whitney U-test for continuous variables. The p-values will be provided for descriptive purposes and will not be considered to define any formal basis for determining factors to be included in statistical models.

Analysis of the primary efficacy variable and outcomes The primary objective of this study is to evaluate the survival free of allograft rejection and re-transplantation after heart transplantation comparing two preservation methods (NIHP versus SCS).

Time-to-event variables (primary efficacy variable) will be analyzed using the Cox proportional hazard model. The estimated hazards ratio and the corresponding two-sided 95% confidence interval will be provided. A supplemental log-rank test will be performed. Survival function for each treatment group will be estimated by Kaplan-Meier method and the Kaplan-Meier curves will be presented. The frequency and percentage of patients who reach the primary composite endpoint will be provided by treatment group for the population.

Analysis of secondary efficacy, exploratory, and safety variables and outcomes The secondary objects of this study are to test if the new preservation technique (NIHP) is superior to standard preservation technique (SCS) in I/R injury (cTnI and CK-MB), immediate graft function, QoL and severe adverse events. Furthermore we will analyse the postoperative renal function (minimum creatinine clearance, need for CRRT), postoperative liver function (ASAT, ALAT), postoperative pulmonary function (hours in ventilator), SAE, time to no improvement in physical activity, resource utilizations (length of stay, and number of visits to professional healthcare).

Continues variables (cTnI, CK-MB, inotrope score, minimum creatinine clearance, hours of ventilator, physical activity (calorie use), length of stay, and number of visits to professional healthcare, EQ-5D index and EQ VAS) will be analysed using Mann-Witney U-test. Additionally, the baseline value of the corresponding variable may be included as a covariate if appropriate. The estimated treatment effect and the corresponding two-sided 95% confidence interval will be provided.

Binary variables (primary graft dysfunction, LVEF<40%, RVEF<40%, severe adverse events) will be analysed using logistic regression. Additionally, the baseline value of the corresponding variable may be included as a covariate if appropriate. The estimated treatment effect and the corresponding two-sided 95% confidence interval will be provided. EQ-5D descriptive system will be analysed by using χ2-test and Fisher's exact test.

SAFETY The assessment of safety will be based primarily on the frequency of adverse events and laboratory abnormalities. Other safety data will be summarized as appropriate. Laboratory data will be summarized by presenting shift tables using extended normal ranges (baseline to most extreme post-baseline value), by presenting summary statistics of raw data and change from baseline values (mean, medians, standard deviations, ranges). An interim assessment of the initial 10 patients in the intervention group will be performed when all of them has passed 30-days post-transplant or expired.

ELIGIBILITY:
Inclusion Criteria recipient:

* Age ≥18 years
* Signed informed consent form
* Listed for heart transplantation

Exclusion Criteria recipient:

* Previous solid organ transplantation
* Grown-up congenital heart disease (GUCH)
* Kidney failure eGFR<40, calculated by CDK-EPI Creatinine, or ultrafiltration or dialysis or rapidly deteriorating kidney function due to a diagnosed renal disease
* Coagulopathy due to known hepatic disease or heparin induced thrombocytopenia
* Ongoing septicemia defined as positive blood culture (including with a durable VAD)
* Incompatible blood group
* Not able to understand the information provided during the informed consent procedure
* Patients under pre-transplant desensitization protocol
* Short term mechanical support pre-transplant (ECMO)
* Patient diagnosed with Systemic Lupus Erythematous, sarcoidosis or amyloidosis
* Combined organ transplantation candidates
* Patient already consented for another transplant related intervention study

Inclusion criteria donor:

* Age ≤70 years
* Accepted as heart donor by the transplant team (research consent from the donor if required in country)

Exclusion criteria donor:

* Previous sternotomy
* DCD hearts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival free of acute cellular rejection and re-transplantation | One year
  The primary end-point is defined as the difference between the two treatment arms in survival free of acute cellular rejection ≥1R and re-transplantation within one year. Acute cellular rejection assessment is based on post-transplant myocardial biopsy information and standard clinical evaluation.

SECONDARY OUTCOMES:
Quality-of-life pre- and posttransplantation | One year
  The EQ-5D-5L, Wellbeing Instrument (OTSWI), and Perceived Threat of the risk for Graft Rejection (PTGR) instruments will be used. This instrument assesses morbidity, self-care, usual activity, pain, anxiety and depression of patients. The instruments will be completed pre-transplant and at 1, 3, 6, and 12 months visits.
I/R-tissue injury | 72 hours
  Cardiac troponin I and T, and kinase-muscle/brain measured at end of preservation and 6±2, 12±4, 24±6, 36±6, 48±6, and 72±6 hours after cross-clamp release.
Immediate graft dysfunction | 24 hours
  Moderate or severe primary graft dysfunction (PGD) within 24 hours after x-clamp release. PGD is measured and defined according to Kobashigawa.
Intermediate graft function | 21 ±7 days post transplantation
  Difference in cardiac dimensions, cardiac output, local and global myocardial perfusion, and extracellular volume will be examined by cardiac magnet resonance at 21 ±7 days post transplantation with a 1.5 Tesla MR scanner.
Chronicle graft rejection | One year post transplant (11- 15 months)
  The number of subject's developed cardiac allograft vasculopathy (CAV), defined as a change in maximal intimal thickness of > 0.5 mm at a specific site in the coronary tree measured by IVUS/OCT at the one-year visit.
Severe adverse events - Cardiac failure | 30 days
  Cardiac failure is determined as the need for intra-aortic balloon pump (IABP) and/or mechanical circulatory extra corporal support (ECMO) within seven days or need for re-transplantation due to graft failure
Severe adverse events - Acute bleeding | 30 days
  Acute bleeding is defined according to the BARC type IV criteria (>2000 ml/24 h and/or requiring re-operation for bleeding, and/or intracranial bleeding, and/or transfusion of >5 red blood cell concentrates/48 h)
Severe adverse events - Respiratory failure | 30 days
  Respiratory failure is defined as impairment of respiratory function requiring re-intubation, tracheostomy, vvECMO or the inability to discontinue invasive ventilator support within 48 h after CPB due to respiratory issues and not due to sedation issues.
Severe adverse events - Acute kidney failure | 30 days
  Acute kidney failure is defined according to the KDIGO criteria as an increase in serum creatinine of >27 μmol/L within 48 hours or 1.5 times baseline within seven days.
Severe adverse events - Permanent stroke | 30 days
  Permanent stroke is defined as an episode of a computer tomography (CT) verified acute neurological dysfunction to be caused by ischemia or haemorrhage, persisting ≥24 hours or until death.
Severe adverse events - Permanent pacemaker | 30 days
  Permanent pacemaker is defined as need for a permanent pacemaker implantation two weeks after transplantation

OTHER OUTCOMES:
Organ discard rate | 24 hours
  Number of donor heart which was discarded after retrieval to the transplant unit
Resource use | One year
  Length of Stay at Intensive Care Unit (ICU) calculated from time patient arrives into the ICU until the patient is discharged from the ICU. Length of Stay at hospital calculated from date and time of surgery until date and time that the patient is discharged from the hospital. Number of visits to professional healthcare within first year post-transplant.
Costs for organ procurement | 24 hours
  Defined as cost for personality, transportation and equipment
Functional capacity | One year
  Recording the patient's activity. Patient will carry an activity monitor (step gauge, accelerator, calorie meter) for the whole day, except when sleeping. The activity clock will also collect information about the patient's heart rhythm. Patient retains the activity meter throughout the study period.
Renal function | 21±7 days post-transplantation
  Difference in renal perfusion and parenchyma examined by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD, PhD, Principal Investigator — Region Skane
Locations (1):
- Skane University Hospital, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steen S, Paskevicius A, Liao Q, Sjoberg T. Safe orthotopic transplantation of hearts harvested 24 hours after brain death and preserved for 24 hours. Scand Cardiovasc J. 2016 Jun;50(3):193-200. doi: 10.3109/14017431.2016.1154598. Epub 2016 Apr 4. PMID 26882241
- [Background] Nilsson J, Jernryd V, Qin G, Nozohoor S, Goncalves DC, Ragnarsson S, Paskevicius A, Johansson M, Warheim J, Hoglund P, Sjoberg T, Steen S. Non Ischemic Heart Preservation. J Heart Lung Transpl 2018;37:S13-S.
- [Background] Jernryd V, Metzsch C, Andersson B, Nilsson J. Organ Preservation and Reperfusion Influence on Outcome after Heart Transplantation. The Journal of Heart and Lung Transplantation 2016;35:S193-S.
- [Background] Nilsson J, Ohlsson M, Stehlik J, Lund L, Andersson B. Prediction of Primary Graft Dysfunction After Heart Transplantation. J Heart Lung Transpl 2015;34:S35-S.
- [Background] Qin G, Sjoberg T, Liao Q, Sun X, Steen S. Intact endothelial and contractile function of coronary artery after 8 hours of heart preservation. Scand Cardiovasc J. 2016 Oct-Dec;50(5-6):362-366. doi: 10.1080/14017431.2016.1213876. Epub 2016 Aug 3. PMID 27420646
- [Background] Steen S. Preservation of the endothelium in cardiovascular surgery-some practical suggestions--a review. Scand Cardiovasc J. 2001 Oct;35(5):297-301. doi: 10.1080/140174301317116253. No abstract available. PMID 11771819
- [Background] Nilsson J, Jernryd V, Qin G, Paskevicius A, Sjoberg T, Hoglund P, Steen S. Non Ischemic Heart Preservation - Results from the Safety Study. J Heart Lung Transpl 2019;38:S26-S.
- [Background] Steen S, Sjoberg T, Pierre L, Liao Q, Eriksson L, Algotsson L. Transplantation of lungs from a non-heart-beating donor. Lancet. 2001 Mar 17;357(9259):825-9. doi: 10.1016/S0140-6736(00)04195-7. PMID 11265950
- [Background] Nilsson J, Jernryd V, Qin G, Paskevicius A, Metzsch C, Sjoberg T, Steen S. A nonrandomized open-label phase 2 trial of nonischemic heart preservation for human heart transplantation. Nat Commun. 2020 Jun 12;11(1):2976. doi: 10.1038/s41467-020-16782-9. PMID 32532991
- [Derived] Pigot H, Steen S, Nilsson J. Comparing non-ischaemic heart preservation (NIHP) with ischaemic static cold storage of donor hearts in adult cardiac transplantation: study protocol for a randomised controlled trial. BMJ Open. 2025 Jun 25;15(6):e100553. doi: 10.1136/bmjopen-2025-100553. PMID 40562558